CLINICAL TRIAL: NCT02669004
Title: Patient-controlled Intermittent Epidural Bolus Versus Epidural Infusion for Posterior Spinal Fusion After Adolescent Idiopathic Scoliosis
Brief Title: Intermittent Epidural Bolus Versus Epidural Infusion for Posterior Spinal Fusion After Adolescent Idiopathic Scoliosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Mehmet Ali Erdoğan, MD, Associate professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: scoliosis
Record Dates: First submitted 2016-01-27; First posted 2016-01-29 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2016-01

CONDITIONS: Pain
Keywords: Analgesia, Epidural,Pain, Postoperative
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intermittent bolus epidural morphine (Active Comparator): Patients who received epidural morphine with patient- controlled intermittent bolus epidural analgesia (PCIEA) represented Group 1. Epidural catheter was inserted by surgeon under direct visualization at the midpoint of the incision and advanced 5-6 cm cephalad to thoracic 4-5 before surgical closure.
  Patients received morphine 50 µg/kg in 10 mL bolus, lockout time 1 hour, no infusion.
  Interventions: Drug: Intermittent bolus epidural morphine
- Continuous epidural morphine (Active Comparator): epidural morphine with patient- controlled continuous epidural analgesia (PCCEA) represented Group 2. Infusion the following initial setting loading morphine 0.02mg/kg in 8mL, was maintained 0.01 mg/kg continuous infusion 4mL, 0.05 mg/kg 2mL bolus dose. 30 minute lock-out interval. 4 hour limit was 4 mg/kg.
  Interventions: Drug: continuous epidural morphine

INTERVENTIONS:
Drug: Intermittent bolus epidural morphine — morphine given with patient- controlled intermittent bolus epidural, 50 µg/kg in 10 mL bolus, lockout time 1 hour, no infusion
  Other Names: PCIEA; Group 1.
  Arms: Intermittent bolus epidural morphine
Drug: continuous epidural morphine — morphine given with patient- controlled continuous epidural, initial setting loading morphine 0.02mg/kg in 8mL, was maintained 0.01 mg/kg continuous infusion 4mL, 0.05 mg/kg 2mL bolus dose. 30 minute lock-out interval. 4 hour limit was 4 mg/kg.
  Other Names: PCCEA; Group 2.
  Arms: Continuous epidural morphine

SUMMARY:
Patient-controlled Intermittent epidural bolus versus epidural infusion for posterior spinal fusion after adolescent idiopathic scoliosis.

Scoliosis surgery is commonly performed in adolescent due to idiopathic scoliosis. It is reported that the postoperative pain after scoliosis surgery that occurs due to Surgical trauma and severe reflex muscle spasm be severe and excruciating. There are many methods for postoperative pain management. It is used often opioid , paracetamol and non-steroidal anti-inflammatory drug with patient- controlled intravenous analgesia (IV-PCA). In addition; intrathecal opioids, one catheter epidural with intermittent dosing bolus of morphine or continuous infusion (either opioids or local anaesthetics or both), double epidural catheter with continuous infusion and intravenous ketamine infusion were preferred other postoperative pain management models.

Epidural analgesia is accepted procedure with the efficacy and safety profile for postoperative pain management in major orthopedic surgery including scoliosis surgery. Epidural analgesia techniques commonly have been used in continuous infusion of local anesthetics with or without opioid. It was emphasized that there was not adequate data in the literature to provide argument concerning the use of epidural opioids after spinal surgery. The objective of this study was to compare the effects and side effects patient- controlled intermittent bolus epidural analgesia (PCIEA) and patient- controlled continuous epidural analgesia (PCCEA) with morphine for postoperative pain control in adolescent idiopathic scoliosis after posterior spinal fusion.

Methods The study was conducted after obtaining written consent from all patients and guardian, approval from the Inonu University Faculty of Medicine Ethics Committee. This prospective randomized controlled double-blinded study was conducted 47 patient between 8-18 years, American Society of Anesthesia Classification (ASA) I-II, with idiopathic scoliosis, scheduled for elective posterior spinal fusion.

Patients with a history of allergy to the drugs used in the study protocol, drug abused , preoperative neurologic deficit, inability to use a visual analogue scale, pulmonary, cardiac and neuropsychiatric disorders were excluded. Exclusion criteria during the study were accidental perforation of dura, faulty epidural catheter placement, postoperative neurologic deficit or uncontrollable nausea, vomiting and pruritus.

The patients who were not premedicated were instructed on the visual analog scale (VAS) and the patient-controlled analgesia (PCA) device that was implanted during the postoperative period.

Patients were divided into two groups using the envelope drawing method. Patients who received epidural morphine with PCIEA represented Group 1, epidural morphine with PCCEA represented Group 2. The anesthetist who collected data and the patients were blinded.

All operations were performed by the same surgical team. The posterior instrumentation with pedicle screws was applied to thoracic and lumbar spine. Epidural catheter was inserted by surgeon under direct visualization at the midpoint of the incision and advanced 5-6 cm cephalad to thoracic 4-5 before surgical closure. Intubated patients was taken to in the reanimation intensive care unit after operation, IV acetaminophen 15 mg / kg was started before extubation and repeated every 6 hours.

After extubation and a neurological examination, patients in the PCİEA group received morphine 50 µg/kg in 10 mL bolus, lockout time 1 hour, no infusion. In Group 2, PCECA infusion the following initial setting loading morphine 0.02mg/kg in 8mL, was maintained 0.01 mg/kg continuous infusion 4mL, 0.05 mg/kg 2mL bolus dose. 30 minute lock-out interval. 4 hour limit was 4 mg/kg.

Pain score, morphine usage, postoperative nausea and vomiting, pruritus, rate their satisfaction ,sedation scores and motor block were assessed by researchers who were blinded to the study groups at postoperatively 2., 4., 6., 8., 12., 18., ve 24.hour, in all patients.

DETAILED DESCRIPTION:
Scoliosis surgery is reported that the postoperative pain after scoliosis surgery that occurs due to Surgical trauma and severe reflex muscle spasm be severe and excruciating. There are many methods for postoperative pain management as opioid , paracetamol and non-steroidal anti-inflammatory drug with patient- controlled intravenous analgesia (IV-PCA). In addition; intrathecal opioids, one catheter epidural with intermittent dosing bolus of morphine or continuous infusion (either opioids or local anaesthetics or both), double epidural catheter with continuous infusion and intravenous ketamine infusion were preferred other postoperative pain management models.

Epidural analgesia is accepted procedure with the efficacy and safety profile for postoperative pain management in major orthopedic surgery including scoliosis surgery. Epidural analgesia techniques commonly have been used in continuous infusion of local anesthetics with or without opioid. It was emphasized that there was not adequate data in the literature to provide argument concerning the use of epidural opioids after spinal surgery. The objective of this study was to compare the effects and side effects patient- controlled intermittent bolus epidural analgesia (PCIEA) and patient- controlled continuous epidural analgesia (PCCEA) with morphine for postoperative pain control in adolescent idiopathic scoliosis after posterior spinal fusion.

Methods This prospective randomized controlled double-blinded study was conducted 47 patient between 8-18 years, American Society of Anesthesia Classification (ASA) I-II, with idiopathic scoliosis, scheduled for elective posterior spinal fusion.

Patients with a history of allergy to the drugs used in the study protocol, drug abused , preoperative neurologic deficit, inability to use a visual analogue scale, pulmonary, cardiac and neuropsychiatric disorders were excluded. Exclusion criteria during the study were accidental perforation of dura, faulty epidural catheter placement, postoperative neurologic deficit or uncontrollable nausea, vomiting and pruritus.

Patients were divided into two groups using the envelope drawing method. Patients who received epidural morphine with PCIEA represented Group 1, epidural morphine with PCCEA represented Group 2. The anesthetist who collected data and the patients were blinded.

All operations were performed by the same surgical team. The posterior instrumentation with pedicle screws was applied to thoracic and lumbar spine. Epidural catheter was inserted by surgeon under direct visualization at the midpoint of the incision and advanced 5-6 cm cephalad to thoracic 4-5 before surgical closure. Intubated patients was taken to in the reanimation intensive care unit after operation, IV acetaminophen 15 mg / kg was started before extubation and repeated every 6 hours.

After extubation and a neurological examination, patients in the PCİEA group received morphine 50 µg/kg in 10 mL bolus, lockout time 1 hour, no infusion. In Group 2, PCECA infusion the following initial setting loading morphine 0.02mg/kg in 8mL, was maintained 0.01 mg/kg continuous infusion 4mL, 0.05 mg/kg 2mL bolus dose. 30 minute lock-out interval. 4 hour limit was 4 mg/kg.

Pain score, morphine usage, postoperative nausea and vomiting, pruritus, rate their satisfaction ,sedation scores and motor block were assessed by researchers who were blinded to the study groups at postoperatively 2., 4., 6., 8., 12., 18., ve 24.hour, in all patients.

The data were given as median with min and max values Statistical analysis was performed using IBM SPSS statistics software 22.0. the groups were compared using Yates' corrected chi-square test and Mann-Whitney U test. Statistical significance was defined as P< 0.05

ELIGIBILITY:
Inclusion Criteria:Clinical diagnosis of idiopathic scoliosis

* scheduled for elective posterior spinal fusion
* American Society of Anesthesia Classification (ASA) I-II

Exclusion Criteria:

* with a history of allergy to the drugs used in the study protocol,
* drug abused ,
* preoperative neurologic deficit,
* inability to use a visual analogue scale, pulmonary,
* cardiac and neuropsychiatric disorders were excluded.

Exclusion criteria during the study:

* accidental perforation of dura,
* faulty epidural catheter placement, postoperative neurologic deficit
* uncontrollable nausea, vomiting and pruritus.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Pain Scores (at movement and at rest) | Postoperatively at 24 hours
  Pain scores were assessed using a visual analog scale (0: No pain, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10: Excruciating pain).

CONTACTS AND LOCATIONS:
Overall Officials: Mahmut Durmuş, Profoser, Study Chair — Inonu University
Locations (1):
- Inonu university, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taenzer AH, Clark C. Efficacy of postoperative epidural analgesia in adolescent scoliosis surgery: a meta-analysis. Paediatr Anaesth. 2010 Feb;20(2):135-43. doi: 10.1111/j.1460-9592.2009.03226.x. PMID 20091934
- [Background] Borgeat A, Blumenthal S. Postoperative pain management following scoliosis surgery. Curr Opin Anaesthesiol. 2008 Jun;21(3):313-6. doi: 10.1097/ACO.0b013e3282f82baa. PMID 18458547
- [Background] Gauger VT, Voepel-Lewis TD, Burke CN, Kostrzewa AJ, Caird MS, Wagner DS, Farley FA. Epidural analgesia compared with intravenous analgesia after pediatric posterior spinal fusion. J Pediatr Orthop. 2009 Sep;29(6):588-93. doi: 10.1097/BPO.0b013e3181b2ba08. PMID 19700988